CLINICAL TRIAL: NCT01488981
Title: A Feasibility Study to Assess the Safety and Efficacy of the Radio-Frequency Microstimulator System to Improve Function of the Arm Following Traumatic Brain Injury
Brief Title: Feasibility of the Radio-Frequency Microstimulator System to Improve Arm Function Following Traumatic Brain Injury
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low enrollment
Sponsor: The Alfred E. Mann Foundation for Scientific Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CP-0014
Record Dates: First submitted 2011-12-05; First posted 2011-12-09 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Traumatic Brain Injury
Keywords: Radio Frequency Microstimulator; Traumatic Brain Injury; TBI; Arm Rehabilitation; electrical stimulation; FES
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Occupational Therapy; Drug Delivery Systems; Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Upper Extremity Therapy without stimulation — Two 12 week phases of occupational therapy without electrical stimulation.
  Other Names: Arm Rehabilitation; Upper Extremity Rehabilitation; Occupational Therapy; OT
Device: Upper Extremity Therapy with stimulation from the Radiofrequency Microstimulator (RFM) System (Alfred Mann Foundation, Santa Clarita, CA) — Two 12 week phases of occupational therapy that incorporates electrical stimulation from the RFM System.
  Other Names: FES; functional electrical stimulation; electrical stimulation

SUMMARY:
This study will evaluate the feasibility of using fully implanted microstimulators to rehabilitate arm function in patients who have suffered a traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) could involve damage to motor pathways within the central nervous system, resulting in loss of arm function from symptoms including general weakness, loss of power, motor control abnormalities and spasticity.

The Radiofrequency Microstimulator (RFM) System consists of fully implanted, leadless stimulators that are injected in a minimally invasive procedure. RFMs measure 16.7mm long, 2.4mm dia. and can be placed directly at target nerves in the arm to drive specific muscle contractions. This system has demonstrated efficacy in arm rehabilitation for stroke patients who suffer from loss of arm function similar to that experienced by some TBI patients.

This feasibility study will evaluate if the RFM system can be used to assist patients in the rehabilitation of arm function following TBI. TBI patients that pass screening will have up to 7 RFM devices implanted in their disabled arm. After implantation, patients will participate in four phases of therapy, each lasting 12 weeks and consisting of standard occupational therapy occurring at regular intervals at home and in the clinic. In the first phase, therapy will not involve use of the RFM System. In the second phase, occupational therapy will be assisted by electrical stimulation using the RFM System. The third and fourth phases will repeat the therapies of the first and second phases, respectively. Arm function following therapy with RFM stimulation will be compared to arm function after therapy without RFM stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject sustained a Traumatic Brain Injury at least 6 and no more than 48 months prior to time of consenting.
2. As a result of Traumatic Brain Injury, subject has impaired hand function associated with poor control and weakness of wrist and elbow extensors on at least one side.
3. Subject has some preserved control of the arm to be treated as demonstrated by any voluntary movement of fingers and shoulder.
4. Subject has functional, passive Range of Motion at the shoulder, elbow, wrist and finger joints of the arm to be treated.
5. Subject's spasticity has been maximally medically controlled and documented stable without change in medication or therapies for a minimum of one month.
6. Peripheral neuromuscular system is intact as demonstrated by electrophysiologic response to routine clinical nerve conduction studies and electromyography on the arm to be treated.
7. Subject is assigned a level no less than VII on the Rancho Los Amigos Levels of Cognitive Functioning Scale.
8. Subject is fluent in English.
9. Subject or their legally authorized representative has signed an informed consent form.
10. Subject (either male or female) is at least 18 years of age at time of consent.
11. Subject is willing and capable of traveling to the investigational site for study visits outlined in this protocol.
12. In the opinion of the Principal Investigator (PI), subject will be able to apply per protocol therapy at home, with the aid of a caregiver if necessary.

Exclusion Criteria:

1. Subject is unwilling to perform all of the therapies and assessments required for the study.
2. Subject has an active implant device (e.g. pacemaker, implanted cardiac defibrillator, neurostimulator, or drug infusion device).
3. Subject has a metal implant (e.g. orthopedic hardware, stent, etc.) that is located within 12 cm of where the RF Coil surface will be placed for the RFM E-Stim therapy.
4. Subject has metal fragments, metal implants, bullet fragments, metal chips or clips in or around the orbits or cranium or any other metal inside the body that would contraindicate an MRI or make it unreadable for the purpose of analysis.
5. Subject with a congenital defect, contracture, upper extremity trauma, or other non-TBI condition that limits range of motion or neuromuscular function of the involved arm.
6. Subject has a documented diagnosis of HIV or other life limiting infection or disease.
7. A female subject who is pregnant, nursing, or planning to become pregnant during the course of the study. Women of childbearing potential must maintain effective contraception during the study period, as judged by the Investigator.
8. Subject has a major psychological disorder, such as poorly controlled schizophrenia or paranoia, such that cooperative status is inconsistent.
9. Subject has severe claustrophobia, movement that cannot be medically controlled or other condition that would limit their ability to undergo an MRI scan or remain still throughout an MRI scan.
10. Subject has non-controlled epilepsy.
11. In the opinion of the PI, subject has a high level of residual spasticity despite maximal medical therapy.
12. Subject has peripheral neuropathy or myopathy in either upper extremity that would preclude implementation of proposed stimulation techniques (i.e. involvement of peripheral nerves or muscles involved in extension of the elbow, wrist, or fingers). An exception is made for carpel tunnel syndrome.
13. Subject has a muscle power grade of more than 3 on the elbow, wrist and finger extensors of the arm to be treated, according to the Medical Research Council (MRC) scale.
14. Subject has a history of endocarditis, a prosthetic valve or murmur.
15. Subject has a history of adverse reactions to anesthetic agents.
16. Recent or current participation in research that may influence response to either study intervention, or be harmful to the subject in any way.
17. Subject's life expectancy is less than 1.5 years.
18. Subject has any bleeding or clotting disorder.
19. Subject has pain that in the opinion of the PI would impair participation.
20. Subject is unwilling to refrain from use of transcutaneous electrical stimulation on the arm to be treated for the duration of their study participation.
21. The PI does not feel the subject is a suitable candidate for the study, for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 2.25 years
  Number of Device-Related Serious Adverse Events during the course of the study.
Action Research Arm Test (ARAT) Score | 12 weeks
  The ARAT is an observational test used to determine upper extremity function. The test measures a subject's ability to perform arm and hand activities of a general nature used in ordinary daily living. These activities are designed to test grasp, pinch, placing, arm extension, elevation, supination and pronation, and, to a lesser extent, strength.
  ARAT score after therapy with RFM stimulation will be compared to ARAT score after therapy without RFM stimulation.

SECONDARY OUTCOMES:
Fugl-Meyer Upper Extremity (FM-UE) Test Score | 12 weeks
  The FM-UE test is an impairment-based Likert scale to assess motor deficits of the upper extremity in neurological patients.
  FM-UE test score after therapy with RFM stimulation will be compared to FM-UE test score after therapy without RFM stimulation.
Wolf Motor Function Test (WMFT) Score | 12 weeks
  The WMFT is a lab-based test focusing on arm function that involves 15 functional tasks and 2 force-based measures which progress in complexity from engaging individual joints to use of the total arm.
  WMFT score after therapy with RFM stimulation will be compared to WMFT score after therapy without RFM stimulation.
Box and Block Test (BBT)Score | 12 weeks
  The BBT measures unilateral gross manual dexterity. The BBT is composed of a wooden box divided in two compartments and 150 blocks. The subject is asked to move as many blocks as possible from one compartment of a box to another, within 60 seconds.
  The number of blocks moved after therapy with RFM stimulation will be compared to the number of blocks moved after therapy without RFM stimulation.
Motor Activity Log (MAL) Score | 12 weeks
  The MAL is a semi-structured interview in which subjects are asked to rate how often they use their impaired arm to complete Activities of Daily Living and how well they are able to complete each Activity.
  MAL score after therapy with RFM stimulation will be compared to MAL score after therapy without RFM stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Subhra Jit Mookerjee, DO, Principal Investigator — James A. Haley VA Medical Center
Locations (1):
- James A. Haley VA Medical Center, Tampa, Florida, United States

REFERENCES:
- See also: Related Info — http://aemf.org